CLINICAL TRIAL: NCT02920593
Title: A Randomized Control Trial of Vitamin D Prophylaxis in the Prevention of Hypertensive Disorders of Pregnancy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Stony Brook University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 875799-3
Record Dates: First submitted 2016-09-09; First posted 2016-09-30 (Estimated); Last update posted 2017-10-05 (Actual); Status verified 2017-10

CONDITIONS: Gestational Hypertension; Toxemia; Superimposed Preeclampsia; Eclampsia; HELLP Syndrome
Keywords: Vitamin D; hypertensive disorders of pregnancy
MeSH Terms: conditions — Hypertension, Pregnancy-Induced; Toxemia; Eclampsia; HELLP Syndrome | interventions — Cholecalciferol; Vitamin D

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Vitamin D Prophylaxis (Experimental): Participants will be provided Vitamin D 3000 IU daily or Vitamin D 4000 IU daily with and without concurrent use of prenatal vitamins, respectively.
  Interventions: Drug: Vitamin D3
- No Vitamin D Prophylaxis (No Intervention): Participants will not receive additional Vitamin D in the pregnancy.

INTERVENTIONS:
Drug: Vitamin D3 — Vitamin D prophylaxis
  Other Names: Vitamin D
  Arms: Vitamin D Prophylaxis

SUMMARY:
The investigators aim to determine if Vitamin D prophylaxis in pregnancy reduces the incidence of hypertensive disorders of pregnancy.

DETAILED DESCRIPTION:
Optimizing Vitamin D status during pregnancy it thought to have maternal, fetal, and neonatal benefit. Studies suggest that Vitamin D acts well beyond its most commonly thought of role in establishing calcium homeostasis and maintaining maternal and neonatal skeletal integrity. Vitamin D has also been found to modulate the maternal renal renin-angiotensin system, maternal immune response, placental implantation and function, and angiogenesis. In light of this, it is no surprise that the 2010 systematic review of vitamin D in pregnancy suggested that Vitamin D deficiency may be associated with an increase risk in maternal and neonatal morbidity. For example, vitamin D deficiency has correlated with an array of maternal conditions, including gestational hypertension, preeclampsia, gestational diabetes, myopathy, vaginal infection, and mental disease. Associated neonatal risks include preterm birth, immunosuppression, infection, low birth weight, hypokalemia, neonatal seizures, asthma, fractures and rickets.

Unfortunately, Vitamin D deficiency in pregnancy is an ongoing epidemic, affecting as many as 82% of pregnant women. While studies on Vitamin D supplementation in pregnancy have consistently shown an associated increase in maternal and neonatal serum Vitamin D levels, some studies have also suggested a concurrent decrease in adverse maternal and neonatal outcomes. For example, Vitamin D supplementation in pregnancies with known deficiency has been shown to decrease the incidence of preeclampsia as much as 32%. Other studies, on the other hand, have suggested no benefit. The inconsistency in findings lie in the fact that these studies were primarily observational in nature and plagued by small sample sizes, recall bias, and inability to adjust for potential confounders. Given this, interpretation regarding clinical significance is limited, preventing providers from making appropriate recommendations to their patients. As such, the American Congress of Obstetricians and Gynecologists (ACOG) has called for high quality studies to address whether the use of Vitamin D supplementation beyond that found in prenatal vitamins is beneficial.

In an effort to elucidate the potential benefit of Vitamin D supplementation in an unscreened population, the investigators propose conducting a randomized control trial in which Vitamin D prophylaxis is provided to a cohort of pregnant women regardless of their Vitamin D status. The aims of the study, therefore, are to:

Specific Aim 1: Determine if Vitamin D prophylaxis in pregnant women decreases the incidence of hypertensive disorders of pregnancy.

Specific Aim 2: Compare neonatal outcomes in those who received Vitamin D prophylaxis to those who did not receive Vitamin D prophylaxis.

Specific Aim 3: Compare placental histology and inflammatory markers in those who received Vitamin D prophylaxis to those who did not receive Vitamin D prophylaxis.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* With a confirmed intrauterine pregnancy, less than 16 weeks gestation
* Carrying a singleton gestation

Exclusion Criteria:

* Taking Vitamin D supplementation outside of prenatal vitamins
* Has a known disorder that will affect vitamin D levels (i.e, hyperparathyroidism, mal-absorption disorder, history of gastric bypass surgery, immunocompromised state, maternal use of immune-modulators etc.)
* Carrying a fetus with known aneuploidy or anomaly
* With fetal demise
* Women with chronic diuretic or cardiac medication therapy including calcium channel blockers

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 412 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-07-31 (Estimated); Study Completion 2019-03-31 (Estimated)

PRIMARY OUTCOMES:
Vitamin D prophylaxis in pregnant women and incidence of hypertensive disorders of pregnancy | 1.5 years
  Number of participants diagnosed with a hypertensive disorder of pregnancy defined as: elevated blood pressure (systolic/diastolic > 140/90mmHg, 2 determinations, 4 hours apart) more than 20 weeks gestation +/- new onset proteinuria (300mg/24hour; protein/creatinine ratio > 3.0mg/dL; 1+ protein on dipstick) or abnormal labs (thrombocytopenia (platelet < 100,000 microliter), impaired liver function testing (AST/ALT twice higher than normal), renal insufficiency (creatinine >1.1mg/dL or doubling of creatinine in the absence of renal disease)) or pulmonary edema or seizure. The outcome will be dichotomized and coded as present or absent.

SECONDARY OUTCOMES:
Adverse neonatal outcome in those who received Vitamin D prophylaxis compared to those who did not receive Vitamin D prophylaxis | 2 years
  The number of participants with an adverse neonatal outcome will be determined by the presence of any of the following pregnancy characteristics: preterm birth <37 weeks; Apgar score <5 at 1 minute, <7 at 5 minutes; low birth weight <2500g; neonatal intensive care unit admission; fetal distress; respiratory distress syndrome; ventilation; neonatal infection; fracture; and neonatal death. The outcome will be dichotomized and coded as present or absent.
Placental pathology in those who received Vitamin D prophylaxis compared to those who did not receive Vitamin D prophylaxis | 2 years
  The number of participants with abnormal placental evaluation will be based on the presence of any of the following: placental abruption, infarction, hypoxia, decidual vasculopathy, or thrombosis of fetal vessels. The outcome will be dichotomized and coded as present or absent.
Placental TNF-alpha in those who received Vitamin D prophylaxis compared to those who did not receive Vitamin D prophylaxis | 2 years
  Number value of placental TNF-alpha level (ng/mL)
Placental inflammatory marker IL-6 in those who received Vitamin D prophylaxis compared to those who did not receive Vitamin D prophylaxis | 2 years
  Number value of placental IL-6 (ng/mL)
Placental inflammatory marker IFN-gamma in those who received Vitamin D prophylaxis compared to those who did not receive Vitamin D prophylaxis | 2 years
  Number value of IFN-gamma (ng/mL)
Placental inflammatory marker GMSCF-2 in those who received Vitamin D prophylaxis compared to those who did not receive Vitamin D prophylaxis | 2 years
  Number value of GMSCF-2 (ng/mL)
Placental inflammatory marker endometrial growth factor in those who received Vitamin D prophylaxis compared to those who did not receive Vitamin D prophylaxis | 2 years
  Number value of endometrial growth factor (ng/mL)
Maternal Vitamin D level in those who received Vitamin D prophylaxis compared to those who did not receive Vitamin D prophylaxis | 1.5 years
  Number value of maternal serum levels of 25(OH)D (ng/mL)
Cord blood Vitamin D level in those who received Vitamin D prophylaxis compared to those who did not receive Vitamin D prophylaxis | 1.5 years
  Number value of cord blood levels of 25(OH)D (ng/mL)

CONTACTS AND LOCATIONS:
Overall Officials: Diana J Garretto, MD, Principal Investigator — SUNY Stony Brook Hospital
Locations (1):
- SUNY Stony Brook Hospital, Stony Brook, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] ACOG Committee Opinion No. 495: Vitamin D: Screening and supplementation during pregnancy. Obstet Gynecol. 2011 Jul;118(1):197-198. doi: 10.1097/AOG.0b013e318227f06b. PMID 21691184
- [Background] Bodnar LM, Catov JM, Simhan HN, Holick MF, Powers RW, Roberts JM. Maternal vitamin D deficiency increases the risk of preeclampsia. J Clin Endocrinol Metab. 2007 Sep;92(9):3517-22. doi: 10.1210/jc.2007-0718. Epub 2007 May 29. PMID 17535985
- [Background] Shin JS, Choi MY, Longtine MS, Nelson DM. Vitamin D effects on pregnancy and the placenta. Placenta. 2010 Dec;31(12):1027-34. doi: 10.1016/j.placenta.2010.08.015. Epub 2010 Sep 22. PMID 20863562
- [Background] Haugen M, Brantsaeter AL, Trogstad L, Alexander J, Roth C, Magnus P, Meltzer HM. Vitamin D supplementation and reduced risk of preeclampsia in nulliparous women. Epidemiology. 2009 Sep;20(5):720-6. doi: 10.1097/EDE.0b013e3181a70f08. PMID 19451820
- [Background] Urrutia RP, Thorp JM. Vitamin D in pregnancy: current concepts. Curr Opin Obstet Gynecol. 2012 Mar;24(2):57-64. doi: 10.1097/GCO.0b013e3283505ab3. PMID 22327734
- [Background] Hollis BW, Johnson D, Hulsey TC, Ebeling M, Wagner CL. Vitamin D supplementation during pregnancy: double-blind, randomized clinical trial of safety and effectiveness. J Bone Miner Res. 2011 Oct;26(10):2341-57. doi: 10.1002/jbmr.463. Erratum In: J Bone Miner Res. 2011 Dec; 26(12):3001. PMID 21706518
- [Background] Shand AW, Nassar N, Von Dadelszen P, Innis SM, Green TJ. Maternal vitamin D status in pregnancy and adverse pregnancy outcomes in a group at high risk for pre-eclampsia. BJOG. 2010 Dec;117(13):1593-8. doi: 10.1111/j.1471-0528.2010.02742.x. Epub 2010 Oct 13. PMID 21040394
- [Background] Johnson DD, Wagner CL, Hulsey TC, McNeil RB, Ebeling M, Hollis BW. Vitamin D deficiency and insufficiency is common during pregnancy. Am J Perinatol. 2011 Jan;28(1):7-12. doi: 10.1055/s-0030-1262505. Epub 2010 Jul 16. PMID 20640974
- [Background] Ringrose JS, PausJenssen AM, Wilson M, Blanco L, Ward H, Wilson TW. Vitamin D and hypertension in pregnancy. Clin Invest Med. 2011 Jun 1;34(3):E147-54. doi: 10.25011/cim.v34i3.15187. PMID 21631991
- [Background] Powe CE, Seely EW, Rana S, Bhan I, Ecker J, Karumanchi SA, Thadhani R. First trimester vitamin D, vitamin D binding protein, and subsequent preeclampsia. Hypertension. 2010 Oct;56(4):758-63. doi: 10.1161/HYPERTENSIONAHA.110.158238. Epub 2010 Aug 23. PMID 20733087
- [Background] Specker B. Vitamin D requirements during pregnancy. Am J Clin Nutr. 2004 Dec;80(6 Suppl):1740S-7S. doi: 10.1093/ajcn/80.6.1740S. PMID 15585798
- [Background] Burton GJ, Sebire NJ, Myatt L, Tannetta D, Wang YL, Sadovsky Y, Staff AC, Redman CW. Optimising sample collection for placental research. Placenta. 2014 Jan;35(1):9-22. doi: 10.1016/j.placenta.2013.11.005. Epub 2013 Nov 19. PMID 24290528
- [Background] Liu NQ, Kaplan AT, Lagishetty V, Ouyang YB, Ouyang Y, Simmons CF, Equils O, Hewison M. Vitamin D and the regulation of placental inflammation. J Immunol. 2011 May 15;186(10):5968-74. doi: 10.4049/jimmunol.1003332. Epub 2011 Apr 11. PMID 21482732
- [Background] Androutsopoulos G, Gkogkos P, Decavalas G. Mid-trimester maternal serum HCG and alpha fetal protein levels: clinical significance and prediction of adverse pregnancy outcome. Int J Endocrinol Metab. 2013 Spring;11(2):102-6. doi: 10.5812/ijem.5014. Epub 2013 Apr 1. PMID 23825981
- [Background] Ertl R, Yu CK, Samaha R, Akolekar R, Nicolaides KH. Maternal serum vitamin D at 11-13 weeks in pregnancies delivering small for gestational age neonates. Fetal Diagn Ther. 2012;31(2):103-8. doi: 10.1159/000333810. Epub 2012 Jan 18. PMID 22261570
- [Background] De-Regil LM, Palacios C, Lombardo LK, Pena-Rosas JP. Vitamin D supplementation for women during pregnancy. Cochrane Database Syst Rev. 2016 Jan 14;(1):CD008873. doi: 10.1002/14651858.CD008873.pub3. PMID 26765344
- [Background] Roth DE. Vitamin D supplementation during pregnancy: safety considerations in the design and interpretation of clinical trials. J Perinatol. 2011 Jul;31(7):449-59. doi: 10.1038/jp.2010.203. Epub 2011 Jan 20. PMID 21252966